CLINICAL TRIAL: NCT03890211
Title: Stepped Wedge Randomized Control Trial of a Non Electric Infant Warmer for Prevention and Treatment of Hypothermia in Rwanda
Brief Title: Trial of a Non Electric Infant Warmer for Prevention and Treatment of Hypothermia in Rwanda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Ministry of Health, Rwanda (Other Government); Rwandan Biomedical Counsel (RBC) (Unknown); Harvard Medical School (HMS and HSDM) (Other); Partners in Health (Other); Rwanda National Ethics Committee (RNEC) (Unknown); Lawrence Berkeley National Laboratory (Unknown)
Responsible Party: Principal Investigator, Anne Hansen, Medical Director of Neonatal Intensive Care Unit, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00030705
Record Dates: First submitted 2019-03-21; First posted 2019-03-26 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Hypothermia Neonatal
Keywords: Hypothermia; Infant Warmer
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Electric Infant Warmer (Experimental): In line with current recommended practice, the mother will be encouraged to provide KMC whenever possible. For hypothermic infants, if the temperature is not rising by ½°C per hour with KMC alone, the Infant Warmer will be offered as an addition. In these cases, the heat will be provided by placing the Infant Warmer over the infant's back while the mother provides KMC. If the mother is not available for KMC at any time, the infant will be warmed exclusively with the Infant Warmer by being placed directly on the warmer as it lies flat. Use of hat and socks will be encouraged by additional clothes will only be added in addition to the warmer per caregiver request, as it reduces heat transfer.
  Interventions: Device: Non-Electric Infant Warmer
- Control (No Intervention): Data such as infant temperature, date of birth, etc. will be collected from those who enroll in the control group. No experimental intervention will be administered.

INTERVENTIONS:
Device: Non-Electric Infant Warmer — Electric warmers are the standard of care in developed countries, but are extremely costly, complicated with risk of causing both hypo and hyperthermia with misuse, and often not feasible in settings without stable electricity. Through a multi-institutional collaboration, the investigators have developed an electricity-free infant warmer.
  Arms: Non-Electric Infant Warmer

SUMMARY:
Hypothermia contributes to a significant portion of neonatal deaths. Kangaroo Mother Care (KMC) is a safe and effective method of warming; however, it is not always feasible, for example in settings such as resuscitation or clinical instability. Electric warmers are the standard of care in developed countries, but are extremely costly, complicated with risk of causing both hypo and hyperthermia with misuse, and often not reliable in settings without stable electricity. After two encouraging pilot studies totaling 204 uses in 2 district hospitals and 4 health centers in rural Rwanda, the investigators aim to further study the warmer in a stepped wedge prospective controlled trial in hospital setting to assess safety and efficacy of the Infant Warmer based on clinical observation and feasibility based on observer audits.

DETAILED DESCRIPTION:
Hypothermia contributes to a significant portion of neonatal deaths. Kangaroo Mother Care (KMC) is a safe and effective method of warming; however, it is not always feasible, for example in settings such as resuscitation or clinical instability. Electric warmers are the standard of care in developed countries, but are extremely costly, complicated with risk of causing both hypo and hyperthermia with misuse, and often not reliable in settings without stable electricity. The Infant Warmer the investigators propose to study has previously been tested in 2 pilot studies totaling 204 uses, occurring in 2 district hospitals and 4 health centers in rural Rwanda.

The combined results of these pilot studies were extremely encouraging. This study will be a stepped wedge prospective controlled trial in hospital setting to assess safety and efficacy of the Infant Warmer based on clinical observation, and feasibility based on observer audits. A total of 10 district hospitals will participate in the study. All 10 hospitals will start with a 2 week period of observation in which "pre" data will be collected. Hospitals will then receive the warmer and be transitioned to the "post" period at a rate of one every two weeks. The primary study aim is to assess the safety, efficacy and feasibility of the Infant Warmer as an addition to KMC, and to achieve and maintain euthermia when KMC is inadequate or unavailable. The study will be conducted across a wide range of district hospitals with control data coming from pre-intervention period and treatment data coming from post intervention period, with the intervention being the introduction of the Infant Warmer.

ELIGIBILITY:
Inclusion Criteria:

Any infant with the following criteria for whom caregiver not available for KMC, or KMC is not adequate (less than 0.5°C/hour rise in temperature):

1. Axillary temperature < 36.5 °C

   a) If an electric warmer is available and the infant's temperature is < 35°C, then the infant will start by being warmed on the electric warmer until the infant's temperature reaches 36°C, then can start non-electric Infant Warmer use.
2. Infants at-risk for hypothermia (criteria: estimated post-menstrual age of < 35 weeks or current body weight of < 2.5 kg).

Exclusion Criteria:

1. Any infant whose family is unwilling to consent to the study.
2. Mothers who are critically ill at the time of infant eligibility or deemed not medically stable by nursing staff to be approached for consent.
3. Any infant with a contraindication to KMC (medical instability) and electrical heating source available.
4. Any infant with initial temperature < 35°C and electrical heating source available.
5. Infants requiring phototherapy.
6. Infants with significant skin condition.

Stop Criteria:

If an electric heating source is available, the infant will be taken off of the study and warmed with an appropriate source of electric heat if the infant:

1. If an electric heating source is available, the infant will be taken off of the study and warmed with an appropriate source of electric heat if the infant:

   i. Has temp < 36 °C while receiving maximum non-electric heat exposure and temperature decreases on any measurement ii. Has temp < 36 °C while receiving maximum non-electric heat exposure and temperature does not begin to rise within 30 minutes iii.Has temp < 36 °C while receiving maximum non-electric heat exposure and not heating at a rate of > ½ °C per hour until temperature >36.5°C iv.Has a temperature that falls below 36°C despite maximum non-electric heat exposure

   Definition of maximum non-electric heat exposure:
   1. IW, KMC, hat; if KMC available
   2. IW, blanket, hat; if KMC not available
   3. Blanket, hat; while seeking caregiver for KMC and/or preparing IW if KMC and IW not available
2. Has temperature > 37.5 °C
3. Is ever considered to be too severely ill by the medical team to be safely cared for in the non-electric Infant Warmer.
4. The warmer will be removed once its temperature drops below phase change temperature as assessed by noting that the material begins to harden and turn white and is no longer warm in area under where baby is lying.

Ages: 0 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3179 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-07-19 (Actual); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Ability to regulate infant body temperature | up to 6 months
  The infant warmer will be evaluated on its ability to achieve and maintain a normal body temperature for patients who are hypothermic and those patients at risk of hypothermia because of a < 2.5 kg birth weight or < 35 week gestational age. Infants temperature will be measured, using a thermometer to ensure the body temperature will increase but not exceed 37.5°C.
Incidence of adverse events as assessed by staff observation | up to 6 months
  The investigators will assess the safety of the infant warmer by observing any adverse reactions such as skin irritations or higher than usual patient temperature (>37.5°C). The safety of the warmer will be measured by study staff observation, measuring the temperature of the warmer with a thermistor instrument, measuring the infant's temperature with a thermometer, as well an investigator-developed Observer Audit Form. The Observer Audit Form is a battery of nine questions which includes eight yes/no questions and one free response. The questions evaluate such topics as whether the warmer was cleaned, the infant was positioned correctly, if adverse events were present, etc.

SECONDARY OUTCOMES:
Studying the practicality of applying the device in a clinical setting | up to 6 months
  The investigators will use observation to evaluate the usability of the warmer by assessing the way that the infant is placed on the warmer and any adverse effects of infant warmer use. This will be measured by study staff observation as well an investigator-developed Observer Audit Form. The Observer Audit Form is a battery of nine questions which includes eight yes/no questions and one free response. The questions evaluate such topics as whether the warmer was cleaned, the infant was positioned correctly, if adverse events were present, etc.
Functionality | up to 6 months
  The functionality will be assessed by the way that the warmer is prepared and cleaned, as well as any wear and tear on the warmer based on repeated use. Functionality will be measured by study staff observation as well an investigator-developed Observer Audit Form. The Observer Audit Form is a battery of eight questions which includes seven yes/no questions and one free response. The questions evaluate such topics as whether the warmer was cleaned, the infant was positioned correctly, if adverse events were present, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Hansen, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Dr Evrard Nahimana, Rwinkwavu, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uwamariya J, Mazimpaka C, May L, Nshimyiryo A, Feldman HA, Sayinzoga F, Umutesi S, Gadgil A, Rapp VH, Nahimana E, Hansen A. Safety and effectiveness of a non-electric infant warmer for hypothermia in Rwanda: A cluster-randomized stepped-wedge trial. EClinicalMedicine. 2021 Apr 16;34:100842. doi: 10.1016/j.eclinm.2021.100842. eCollection 2021 Apr. PMID 33997734